CLINICAL TRIAL: NCT06005129
Title: Engaging Higher-Order Mechanisms of Psychopathology: A Parsimonious Approach to Precision Medicine
Brief Title: Personality Change Study for Borderline Personality Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shannon E. Sauer-Zavala (Other)
Collaborators: American Psychological Foundation (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Shannon E. Sauer-Zavala, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 86801; R61MH133665 (NIH)
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personality-based treatment 2 week baseline (Experimental): Participants will receive treatment tailored to 1 of 3 personality dimensions after a 2 week baseline assessment
  Interventions: Behavioral: Personality-Based Therapy
- Personality-based treatment 4 week baseline (Experimental): Participants will receive treatment tailored to 1 of 3 personality dimensions after a 4 week baseline assessment
  Interventions: Behavioral: Personality-Based Therapy

INTERVENTIONS:
Behavioral: Personality-Based Therapy — Participants will be randomized to a 2- or 4-week assessment-only baseline period. After the baseline period, participants will receive the personality-based treatment module corresponding to their highest clinical elevation (i.e., neuroticism, [low] conscientiousness, [low] agreeableness). Treatment will consist of six weekly 50-60-minute sessions. After the 6-week intervention period, participants will complete a 4-week follow-up period to determine the sustainability of effects observed

SUMMARY:
Participants with borderline personality disorder will undergo an a 2 - 4 week baseline assessment to determine level of outcomes of interest in the absence of treatment. After the baseline period, participants will receive six weekly 50-60-minute treatment sessions. After the 6 treatment sessions, participants will complete a 4-week follow-up period to determine the sustainability of the treatment module.

ELIGIBILITY:
Inclusion Criteria:

* Speak English fluently
* Diagnosis of Borderline Personality Disorder

Exclusion Criteria:

* diagnosed psychological conditions that would be better addressed by alternative treatments
* concurrent psychotherapy
* medication instability
* substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in clinician-rated borderline personality disorder symptoms | up to 14 weeks (pre-baseline, pre-intervention, post-intervention, post-follow-up)
  Change in borderline personality disorder symptoms will be measured using Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) - clinician-rated version. Scores range from 0-36; higher scores indicate greater severity of borderline personality disorder symptoms
Change in patient-reported borderline personality disorder symptoms | weekly up to 14 weeks
  Change in borderline personality disorder symptoms will be measured using Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) - self-report version. Scores range from 0-36; higher scores indicate greater severity of borderline personality disorder symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Sauer-Zavala, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Clinic for Emotional Health at the University of Kentucky, Lexington, Kentucky, United States